CLINICAL TRIAL: NCT06725056
Title: Detachable String Magnetically Controlled Capsule Endoscopy for Patients with Acute Upper Gastrointestinal Bleeding: a Prospective Study
Brief Title: Detachable String Magnetically Controlled Capsule Endoscopy for Patients with AUGIB
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhuan Liao, Professor, Changhai Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: DS-MCE for patients with AUGIB
Record Dates: First submitted 2024-10-19; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Acute Upper Gastrointestinal Bleeding; Capsule Endoscopes
Keywords: AUGIB; DS-MCE; emergency department
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- group of participants (Experimental): Sequentially performing DS-MCE and EGD examinations on AUGIB patients with stable hemodynamics, using EGD as the gold standard to evaluate the sensitivity of DS-MCE in diagnosing upper gastrointestinal bleeding lesions and active bleeding.
  Interventions: Other: DS-MCE and EGD examinations

INTERVENTIONS:
Other: DS-MCE and EGD examinations — sequentially performing DS-MCE and EGD examinations on AUGIB patients with stable hemodynamics

SUMMARY:
Use CE for pre-examination of patients with AUGIB symptoms in emergency centers may reduce the need for emergency electronic gastroscopy and have certain advantages in clinical work. Patients with low-risk lesions can be discharged without the need for EGD and hospitalization, greatly improving the utilization of medical resources.

DETAILED DESCRIPTION:
The investigators plan to conduct exploratory research by sequentially performing DS-MCE and EGD examinations on AUGIB patients with stable hemodynamics, using EGD as the gold standard to evaluate the sensitivity of DS-MCE in diagnosing upper gastrointestinal bleeding lesions and active bleeding.

ELIGIBILITY:
Inclusion Criteria:

* No gender limit, age ≥ 18 years
* Presenting to the emergency department with melena or hematemesis
* Hemodynamically stable at presentation
* No endoscopic examination has been performed due to this bleeding
* Agree to participate in this clinical trial and sign an informed consent form

Exclusion Criteria:

* Patients with acute active massive bleeding or hemodynamic instability (blood pressure < 90 mmHg and heart rate > 120 beats per minute)
* Patients with Hematochezia
* Hemodynamics remained unstable after fluid resuscitation
* Known or suspected intestinal obstruction, stenosis, or fistula
* Severe motor disorders such as asthma, swallowing disorders, or gastric paralysis
* History of abdominal surgery that affects the normal structure of the digestive tract in the past
* When capsule retention occurs, the problem cannot be solved through surgery due to subjective or objective reasons
* Implantable medical devices such as pacemakers, electronic cochlear implants, drug infusion pumps, and neural stimulators are installed inside the body, except for MRI compatible products
* Pregnant women
* Those who require MRI examination before capsule endoscopy discharge
* Suffering from severe cardiovascular and pulmonary diseases (such as severe myocardial infarction, arrhythmia, heart failure, and respiratory failure)
* Refuse MCE or gastroscopy examination
* The researchers believe that the subjects have any other factors that are not suitable for participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-25 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity of DS-MCE in detection active bleeding and bleeding lesions, using the detection of EGD as the gold standard, | From enrollment to the end of end of follow-up at 4 weeks
  Active bleeding is defined as the continuous flow of visible blood from damaged blood vessels under the microscope.
  The detection results of bleeding lesions are divided into three categories: P0 refers to lesions without possible bleeding, such as visible submucosal veins, diverticula without bleeding traces, nodules without mucosal damage traces, etc; P1 refers to low-risk bleeding lesions, such as isolated erythema, isolated small erosions, or mucosal damage; P2 refers to high-risk bleeding lesions, such as peptic ulcers (active bleeding or visible blood vessels) with persistent or rebleeding risks, erosions with a diameter of ≥ 2mm, tumors, varicose veins, etc.

SECONDARY OUTCOMES:
The specificity of ds MCE in detecting active bleeding and bleeding lesions using EGD as the gold standard | From enrollment to the end of end of follow-up at 4 weeks
The number of observed signs of bleeding | From enrollment to the end of end of follow-up at 4 weeks
Detection rate of bleeding lesions in enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
Detection rate of lesions in enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
The time from the admission of subjects to the detection of bleeding lesions | From enrollment to the end of end of follow-up at 4 weeks
Number of therapeutic interventions (endoscopy, DSA, surgery) for enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
The time from the admission of subjects to the start of therapeutic interventions (endoscopy, DSA, surgery) | From enrollment to the end of end of follow-up at 4 weeks
Detection rate of esophageal, gastric, and small intestinal lesions in enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
Time of traditional electronic gastroscopy examination | From enrollment to the end of end of follow-up at 4 weeks
Time of DS-MCE examination | From enrollment to the end of end of follow-up at 4 weeks
Incidence of rebleeding in enrolled subjects 30 days after discharge | From enrollment to the end of end of follow-up at 4 weeks
Rate of all-cause mortality among enrolled subjects within 30 days of discharge | From enrollment to the end of end of follow-up at 4 weeks
Time of hospital stay for enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
Satisfaction of enrolled subjects | From enrollment to the end of end of follow-up at 4 weeks
  use a certain scale named satisfaction scale to measure the satisfaction of enrolled subjects (0-36), lower scores mean a better outcome.
clinical safety (Incidence of Treatment-Emergent Adverse Events, Safety and Tolerability) | From enrollment to the end of end of follow-up at 4 weeks
  use the incidence of adverse events to measure clinical safety
complication rate | From enrollment to the end of end of follow-up at 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhuan Liao, Study Chair — Changhai Hospital
Locations (1):
- Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No